CLINICAL TRIAL: NCT01846481
Title: A Randomized, Double-blind, Placebo-controlled, Dose of RBP-8000 Following IV Cocaine to Evaluate the Pharmacokinetics Parameters of RBP-8000 and Cocaine and to Assess the Effects of Drug on Cocaine-induced Physiologic and Behavioral Effects in Cocaine Abusing Subjects
Brief Title: A Randomized, 4-sequence, 2-period, Double-blind, Placebo Controlled Study With a DSM-IV-TR Diagnosis of Cocaine Abuse
Acronym: RBP-8000
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Indivior Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RB-US-13-0004
Record Dates: First submitted 2013-05-01; First posted 2013-05-03 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-09

CONDITIONS: Opioid Dependence; Opioid Related Disorders; Cocaine Dependence
Keywords: Cocaine
MeSH Terms: conditions — Opioid-Related Disorders; Cocaine-Related Disorders | interventions — RBP-8000; Cocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- RBP-8000 100mg/Placebo (Experimental): Day 1: 50mg intravenous infusion of cocaine
  Day 3: 50mg intravenous infusion of cocaine followed by a 100mg intravenous infusion of RBP-8000
  Day 6: 50mg intravenous infusion of cocaine followed by an intravenous infusion of placebo
  Interventions: Drug: RBP-8000 100 mg; Drug: Placebo; Drug: Cocaine
- Placebo/RBP-8000 100mg (Experimental): Day 1: 50mg intravenous infusion of cocaine
  Day 3: 50mg intravenous infusion of cocaine followed by an intravenous infusion of placebo
  Day 6: 50mg intravenous infusion of cocaine followed by a 100mg intravenous infusion of RBP-8000
  Interventions: Drug: RBP-8000 100 mg; Drug: Placebo; Drug: Cocaine
- RBP-8000 200mg/Placebo (Experimental): Day 1: 50mg intravenous infusion of cocaine
  Day 3: 50mg intravenous infusion of cocaine followed by a 200mg intravenous infusion of RBP-8000
  Day 6: 50mg intravenous infusion of cocaine followed by an intravenous infusion of placebo
  Interventions: Drug: Placebo; Drug: Cocaine; Drug: RBP-8000 200 mg
- Placebo/RBP-8000 200mg (Experimental): Day 1: 50mg intravenous infusion of cocaine
  Day 3: 50mg intravenous infusion of cocaine followed by an intravenous infusion of placebo
  Day 6: 50mg intravenous infusion of cocaine followed by a 200mg intravenous infusion of RBP-8000
  Interventions: Drug: Placebo; Drug: Cocaine; Drug: RBP-8000 200 mg

INTERVENTIONS:
Drug: RBP-8000 100 mg — RBP-8000 100 mg administered in the vein on either study day 3 or 6. There is a 72-hour washout between Days 3 and 6
  Other Names: T172R/G173G cocaine esterase
  Arms: Placebo/RBP-8000 100mg; RBP-8000 100mg/Placebo
Drug: Placebo — IV infusion of Placebo administered 1 minute after cocaine infusion on either day 3 or 6.
Drug: Cocaine — 50 mg intravenous (IV) dose of cocaine administered over 10 minutes on Days 1, 3 and 6.
  Other Names: Benzoylmethylecgonine
Drug: RBP-8000 200 mg — RBP-8000 200 mg administered in the vein on either study day 3 or 6. There is a 72-hour washout between Days 3 and 6
  Other Names: T172R/G173G cocaine esterase
  Arms: Placebo/RBP-8000 200mg; RBP-8000 200mg/Placebo

SUMMARY:
This is a randomized, 4-sequence, 2-period, double-blind, placebo controlled study in male and female subjects with an American Psychiatric Association Diagnostic and Statistical Manual DSM-IV-TR diagnosis of cocaine abuse.

DETAILED DESCRIPTION:
There will be a 28-day screening period with eligible subjects remaining resident in the clinic from the evening before Day -1 up and until the morning of Day 9. On the morning of Day 1, a 50 mg intravenous (IV) infusion of cocaine will be administered over 10 minutes to all subjects. If none of the stopping criteria were met and no intervening safety concerns, subjects will be randomized to one of the treatment sequences on Day 3. On dosing days, Day 3 and Day 6, subjects will have fasted at least 8 hours before dosing of cocaine and either RBP-8000 200 mg, RBP-8000 100 mg or matching placebo.

ELIGIBILITY:
Inclusion Criteria:

* Male and female volunteers aged 21-50 years, inclusive
* Body mass index (BMI)18-32 kg/m^2 and weight of at least 50 kg
* Not currently seeking treatment for substance abuse or substance dependence
* Subject is healthy, in the opinion of the Principal Investigator other than cocaine abuse; as determined by the absence of clinically significant medical/psychiatric history or findings, particularly cardiovascular or central nervous system (CNS) disease, physical examination, normal renal function, ECG findings, vital signs, and laboratory results at screening
* Males agree to refrain from sperm donations for the entire duration of the study, and for at least 90 days after the last dose of study drug
* Has experience using cocaine by the smoked or IV route at least 6 times in past 12 months and a positive urine drug screen for cocaine prior to study intake (Day -2). Has experience using cocaine by the smoked or IV route in the past 3 months and a positive urine drug screen for cocaine during screening prior to study check-in at the clinic
* Be able to verbalize understanding of the consent form, able to provide written informed consent, and verbalize willingness to complete study procedures, prior to the initiation of any protocol-specific procedures
* Meet DSM-IV-TR criteria for current cocaine abuse
* Be able to comply with protocol requirements, rules, and regulations of the study site, and be likely to complete all the study procedures in the opinion of the Principal Investigator

Exclusion Criteria:

* Current or past history of seizure disorder, including alcohol- and/or stimulant-related seizure, febrile seizure, or significant family history of idiopathic seizure disorder. Have any previous clinically significant reaction to cocaine, including loss of consciousness or seizure
* Current alcohol dependence or current drug dependence according to DSM-IV-TR criteria (excluding nicotine and caffeine)
* Clinically significant history of cardiac disease, including cardiovascular and conduction abnormalities or ECG evidence of cardiac abnormalities
* QTcF greater than or equal to 450 for male subjects and 470 for female subjects as measured through a 12-lead ECG
* History of liver disease or current elevation of aspartate aminotransferase (AST) or alanine aminotransferase (ALT) exceeding 3x the upper limit of normal
* Be on probation or parole, and/or have current or pending legal charges with the potential for incarceration that could interfere with the study scheduling
* Women with a positive pregnancy test at screening; or women who are pregnant or lactating or who are seeking to become pregnant
* Women of childbearing potential (who are sexually active with a male) who fail to use medically acceptable contraception methods (e.g., an oral or injectable contraceptive, an approved hormonal implant or topical patch, an intrauterine device, a double barrier method, or barrier plus spermicide). A woman of childbearing potential is defined as any female who is less than 2 years post-menopausal or has not undergone a hysterectomy or surgical sterilization, e.g., bilateral tubal ligation, bilateral ovariectomy (oophorectomy). Females that are post-menopausal will be confirmed as such by the follicle stimulating hormone (FSH) test at initial screening
* Males who do not agree to use barrier contraception and spermicide when engaging in sexual activity with a female of child-bearing potential while on study medication, and for at least 28 days after the last dose of study medication
* History of clinically significant severe allergic or anaphylactic reactions

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2013-04; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration (Cmax) of Cocaine, (-)Ecgonine methyl ester and RBP-8000 | 21 samples from pre-dose of cocaine up to 731 minutes after start of cocaine infusion
Time to Maximum Plasma Concentration (Tmax) of Cocaine, (-)Ecgonine methyl ester and RBP-8000 | 21 samples from pre-dose of cocaine up to 731 minutes after start of cocaine infusion
Area under the plasma concentration-time curve from time 0 to the last quantifiable concentration (AUClast) of Cocaine, (-)Ecgonine methyl ester and RBP-8000 | 21 samples from pre-dose of cocaine up to 731 minutes after start of cocaine infusion
Elimination half-life (t1/2) of Cocaine, (-)Ecgonine methyl ester and RBP-8000 | 21 samples from pre-dose of cocaine up to 731 minutes after start of cocaine infusion
Area under the plasma concentration-time curve from time 0 to theoretical infinity (AUC0-inf) of Cocaine, (-)Ecgonine methyl ester and RBP-8000 | 21 samples from pre-dose of cocaine up to 731 minutes after start of cocaine infusion
Distribution half-life (t1/2α) of Cocaine | 21 samples from pre-dose of cocaine up to 731 minutes after start of cocaine infusion
Clearance (CL) of Cocaine, (-)Ecgonine methyl ester and RBP-8000 | 21 samples from pre-dose of cocaine up to 731 minutes after start of cocaine infusion
Volume of distribution (Vd) of Cocaine, (-)Ecgonine methyl ester and RBP-8000 | 21 samples from pre-dose of cocaine up to 731 minutes after start of cocaine infusion
Elimination rate constant (λz) of Cocaine, (-)Ecgonine methyl ester and RBP-8000 | 21 samples from pre-dose of cocaine up to 731 minutes after start of cocaine infusion
Mean residence time (MRT) of Cocaine, (-)Ecgonine methyl ester and RBP-8000 | 21 samples from pre-dose of cocaine up to 731 minutes after start of cocaine infusion

SECONDARY OUTCOMES:
Behavioral effects - as Measured by the Participant Using the Brief Substance Craving Scale | Post dosing 30 min,1,0, 2.0, 3.0, 4.0, 7.0, 8.0, 12.0,24.0 hours

CONTACTS AND LOCATIONS:
Overall Officials: Bradley D Vince, DO, Principal Investigator — Vince and Associates Clinical Research
Locations (1):
- Vince and Associates Clinical Research, Overland Park, Kansas, United States